CLINICAL TRIAL: NCT07219706
Title: Examining the Independent and Combined Effects of Dietary Fiber and Time Restricted Eating on Indicators of Cancer Risk: the Fiber and Time Restricted Eating (F.I.T.) Study
Brief Title: Dietary Fiber and Time Restricted Eating
Acronym: FIBER+TRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 18665
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diet Habits; Cancer Prevention
Keywords: Diet; Weight loss; Fasting; Time restricted eating; Time restricted feeding
MeSH Terms: conditions — Feeding Behavior; Weight Loss; Fasting; Intermittent Fasting | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fiber for Improvement of Behavior, Eating, and Risk (FIBER) (Experimental)
  Interventions: Behavioral: Group education; Behavioral: Counseling
- Time Restricted Eating (TRE) (Experimental)
  Interventions: Behavioral: Time Restricted Eating
- FIBER and TRE (Experimental)
  Interventions: Behavioral: Time Restricted Eating; Behavioral: Group education; Behavioral: Counseling

INTERVENTIONS:
Behavioral: Time Restricted Eating — 10-hour Time Restricted Eating (TRE)
  Arms: FIBER and TRE; Time Restricted Eating (TRE)
Behavioral: Group education — Group education about dietary fiber
  Arms: FIBER and TRE; Fiber for Improvement of Behavior, Eating, and Risk (FIBER)
Behavioral: Counseling — Counseling and motivational interviewing to promote uptake of diet changes
  Arms: FIBER and TRE; Fiber for Improvement of Behavior, Eating, and Risk (FIBER)

SUMMARY:
This study is seeking to examine combinations of two different dietary interventions on cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 age
* Body mass index ≥30 kg/m2
* Dietary fiber intake ≤15 g/day
* Compatible cell phone for use of ecological momentary assessment app

Exclusion Criteria:

* Self-reported diagnosis that precludes fiber intake (e.g., inflammatory bowel disease)
* Food allergies or intolerances that limit ability to engage with the intervention
* Positive screen on the SCOFF eating disorder screener39
* Current self-reported use of GLP-1 receptor agonists
* Currently pregnant or breastfeeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Dietary fiber intake | Baseline, post-intervention (approximately 3 months), and post-observation (approximately 12 months)
  Dietary fiber intake as reported on 3-day diet records and analyzed according to Nutrition Data System for Research; reported as a mean intake over three days in grams per day

SECONDARY OUTCOMES:
Body mass/weight | Baseline, post-intervention (approximately 3 months), and post-observation (approximately 12 months)
  Body mass/weight will be measured in kilograms
Blood pressure | Baseline, post-intervention (approximately 3 months), and post-observation (approximately 12 months)
  Blood pressure (systolic and diastolic) will be measured at each time frame (in millimeters of mercury [mmHg])
Blood-based measures of inflammation | Baseline, post-intervention (approximately 3 months), and post-observation (approximately 12 months)
  Venous blood samples will be collected and analyzed for inflammatory markers: Granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon-gamma (IFN-γ), interleukin-1 beta (IL-1β), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), and tumor necrosis factor-alpha (TNF-α).
Blood-based measures of oxidative stress | Baseline, post-intervention (approximately 3 months), and post-observation (approximately 12 months)
  Venous blood samples will be collected and analyzed for measures of oxidative stress, including reactive oxygen species and lipid peroxidation
Blood-based measures of insulin resistance | Baseline, post-intervention (approximately 3 months), and post-observation (approximately 12 months)
  Insulin resistance will be measured via assessment of insulin and glucose in venous blood samples, and used to assess Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Affect | Daily for three months
  Self-reported affect will be assessed using ecological momentary assessment, delivered via cell phone
Sleep | Daily for three months
  Sleep will be measured via Fitbits, assessed as mean minutes/night
Physical Activity | Daily for three months
  Physical activity will be measured via Fitbits, assessed as mean steps/day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No